CLINICAL TRIAL: NCT04261647
Title: The Effect of Adding Kinesio-taping Versus Pelvic Floor Exercise to Conventional Therapy in the Management of Post-colonoscopy Coccydynia
Brief Title: Kinesio-taping Versus Pelvic Floor Exercise for Post Colonoscopy Coccydynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadaya Mosaad (Other)
Responsible Party: Sponsor-Investigator, Hadaya Mosaad, lecturer at physical therapy department for Surgery, Cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012002613
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Musculoskeletal Pain
Keywords: pelvic floor exercise; coccydynia
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): kinesio- taping technique plus traditional physical therapy program.
  Interventions: Other: kinesio-taping techniques.; Other: traditional physical therapy program , stretching of piriformis. iliopsoas, clam shell exercise,seat cushioning and seat kitz.
- Experimental group 2 (Experimental): Pelvic floor exercise plus traditional physical therapy program.
  Interventions: Other: Pelvic floor exercise; Other: traditional physical therapy program , stretching of piriformis. iliopsoas, clam shell exercise,seat cushioning and seat kitz.
- Control group (Active Comparator): traditional physical therapy program in the form of stretching of piriformis, stretching of iliopsoas and clam shell exercise, seat cushioning and seat kitz.
  Interventions: Other: traditional physical therapy program , stretching of piriformis. iliopsoas, clam shell exercise,seat cushioning and seat kitz.

INTERVENTIONS:
Other: kinesio-taping techniques.
  Arms: Experimental group 1
Other: Pelvic floor exercise
  Arms: Experimental group 2
Other: traditional physical therapy program , stretching of piriformis. iliopsoas, clam shell exercise,seat cushioning and seat kitz.

SUMMARY:
Forty-two patients, with coccydynia following colonoscopy were selected from Kasr El-Aini teaching Hospital, with age ranged from 25-45 years. Patients were randomly assigned to the control or experimental groups. The patients in the three groups completed 3-weeks 3 sessions per week for traditional physical therapy treatment consisting of stretching exercise for the piriformis and iliopsoas muscles, clamshell exercise, seat cushioning and seat kitz. Experimental group I received kinsiotaping techniques in addition to the traditional physical therapy. While experimental group II received pelvic floor exercise in the form of reverse kegel exercise or pelvic pulges, in addition to conventional therapies. pain intensity were evaluated by numerical rating scale as a primary out come measure, and Oswestry disability index was used as a secondary out come measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from pain in or around the coccyx, following colonoscopy procedures.
* Age group ranging from 38-58 years old.

Exclusion Criteria:

* Cancer.

  , - Cysts in pelvic area.
* Pelvic fracture or recent trauma.
* Patient with pain in coccyx region referred from lumbar spine, pelvic floor muscles, degenerative disc, neoplasms, bony spurs, or infections.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
pain intensity measured by numerical rating scale. | after 3 weeks of intervention.
  a one-dimensional measure of pain intensity in adults, including those with chronic pain. Numerical pain rating scale consists an 11-point numeric scale with 0 representing "no pain" and 10 representing extreme pain (Worst possible pain)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol statistical analusis.
Supporting Information: Study Protocol, SAP
Time Frame: We will share the results after 6 months from publication.